CLINICAL TRIAL: NCT05735340
Title: Evaluating the Feasibility of Type 1 Diabetes Education and Support Intervention to Improve Diabetes Distress Among Black Young Adults
Brief Title: Type 1 Diabetes Education and Support Study
Acronym: T1DES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RNG211852; 1R01DK128236-01A1 (NIH)
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Type1diabetes
Keywords: diabetes; type 1
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Education (Active Comparator): Participants in this arm will receive traditional diabetes education following a baseline assessment. During months 1-3, participants will attend 5 sessions. Follow-up will be conducted at 3-months and 6-months.
  Interventions: Behavioral: Diabetes Education
- T1DES (Experimental): Participants in this arm will receive a emotion regulation intervention called T1DES following a baseline assessment. During months 1-3, participants will attend 5 sessions. Follow-up will be conducted at 3-months and 6-months.
  Interventions: Behavioral: T1DES

INTERVENTIONS:
Behavioral: Diabetes Education — Participants in this arm will receive traditional diabetes education over 5 sessions in the first 3 months of participation and be followed for 6 months.
  Arms: Diabetes Education
Behavioral: T1DES — Participants in this arm will receive the T1DES behavioral interventions over 5 sessions in the first 3 months of participation and be followed for 6 months.
  Arms: T1DES

SUMMARY:
Diabetes distress has been identified as one of the largest contributors to the racial disparity in glycemic control that disproportionately burdens Black patients ages 18-30 years with type 1 diabetes (T1D). In order to combat this issue, this study assesses the feasibility of the culturally tailored intervention T1DES and evaluates the effect of the T1DES intervention on diabetes outcomes in a pilot randomized clinical trial among Black young adults with T1D.

DETAILED DESCRIPTION:
This research focuses on the unique needs of Black young adults aged 18-30 years to address a critical gap in the research and clinical care. The goal is to test the feasibility and preliminary efficacy of a culturally adapted and tailored intervention to enhance diabetes management strategies among Black young adults with T1D, addressing the pervasive racial disparity in health outcomes for this population.

The specific aims for this study are to:

Aim 1: Assess feasibility of the culturally tailored intervention T1DES by measuring intervention acceptability, demand (retention, completed > 80% of sessions), practicality, and implementation fidelity through participant surveys and key informant interviews with participants and the health care delivery team.

Aim 2: Evaluate the effect of the T1DES intervention on diabetes outcomes in a pilot randomized clinical trial among N=40 Black young adults age 18-30 years with T1D and elevated HbA1c (>7.5%) by comparing changes in HbA1c, diabetes distress, and self-management from baseline to 6-months post-baseline among participants randomized to T1DES compared to the diabetes education-only control condition.

The goal of this study is to provide diabetes education and emotion regulation support tailored for Black young adults' experiences that will result in sustained glycemic control and can be incorporated into adult endocrinology practices.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Georgia Member
* Aged 18 - 30 years
* Confirmed diagnosis of Type 1 diabetes
* Hemoglobin A1c > 7.5 at time of enrollment
* a cell phone able to send/receive text messages
* Self-reported race of Black or African American
* Ability to read in English and provide informed consent

Exclusion Criteria:

* Developmental delay or other cognitive impairment that would render the participant unable to provide informed consent
* Subjects with visual impairment or have severe hearing or other physical disabilities that would be a barrier for participating in-group or web sessions
* Diabetes complications that would preclude participation in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | 3 months
  Problem Areas in Diabetes - Emerging Adults 25 Item Measure and Scoring. Higher scores indicate more diabetes distress, with a range from 0 to 100.
Diabetes Distress | 6 months
  Problem Areas in Diabetes - Emerging Adults 25 Item Measure and Scoring. Higher scores indicate more diabetes distress, with a range from 0 to 100.
Diabetes Distress | 3 months
  Type 1 Diabetes Distress Scale. Higher scores indicate more diabetes distress, with a range from 1 to 6.
Diabetes Distress | 6 months
  Type 1 Diabetes Distress Scale. Higher scores indicate more diabetes distress, with a range from 1 to 6.
A1C | 3 months
  Point of Care A1C
A1C | 6months
  Point of Care A1C

CONTACTS AND LOCATIONS:
Overall Officials: Teaniese L Davis, PhD, MPH, Principal Investigator — Principal Investigator
Locations (1):
- Kaiser Permanente Georgia, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No